CLINICAL TRIAL: NCT04671953
Title: An Open-label, Two-arm Crossover Study to Investigate the Effect of BMS-986165 on the Pharmacokinetics of Metformin in Healthy Volunteers
Brief Title: Effect of BMS-986165 on the Blood Levels of Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-159
Record Dates: First submitted 2020-12-15; First posted 2020-12-17 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Healthy Participants
Keywords: Drug interaction; Metformin; Pharmacodynamics; Pharmacokinetics
MeSH Terms: interventions — deucravacitinib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: BMS-986165 Dose 1 + Metformin (Experimental)
  Interventions: Drug: BMS-986165; Drug: Metformin
- Arm 2: BMS-986165 Dose 2 + Metformin (Experimental)
  Interventions: Drug: BMS-986165; Drug: Metformin

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Other Names: Deucravacitinib
Drug: Metformin — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate the effects of BMS-986165 on the drug levels of metformin in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy, as determined by having no clinically significant deviation from normal in medical history, physical examination, electrocardiograms, vital signs, and clinical laboratory determinations
* Body mass index of 18.0 kg/m^2 to 32.0 kg/m^2, inclusive, and body weight ≥ 50 kg, at screening
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

- Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) in plasma for metformin with and without BMS-986165 | Up to 9 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC (0-T)) in plasma for metformin with and without BMS-986165 | Up to 9 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) in plasma for metformin with and without BMS-986165 | Up to 9 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 13 days
Incidence of serious adverse events (SAEs) | Up to 71 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 41 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 41 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 41 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 41 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 41 days
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS | Up to 41 days
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 41 days
  The QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF | Up to 41 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in clinical laboratory values: Hematology tests | Up to 41 days
Incidence of clinically significant changes in clinical laboratory values: Clinical chemistry tests | Up to 41 days
Incidence of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 41 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm